CLINICAL TRIAL: NCT00114192
Title: Phase II Study of Docetaxel and Thalidomide as a Second-Line Treatment for Non-Small Cell Lung Cancer
Brief Title: Docetaxel and Thalidomide as Second-Line Therapy in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 11212; UVACC-HIC-11212; UVACC-LUNG3; UVACC-29403
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2010-01

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Thalidomide may stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Thalidomide may also help docetaxel work better by making tumor cells more sensitive to the drug. Giving docetaxel together with thalidomide may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel together with thalidomide works as second-line therapy in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete and partial response rates in patients with stage III or IV non-small cell lung cancer treated with docetaxel and thalidomide as second-line therapy.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the response duration and survival of patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive docetaxel IV over 30-60 minutes on days 1, 8, and 15. Patients also receive oral thalidomide once daily on days -7 to 28 for course 1 and on days 1-28 for all subsequent courses. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease after 6 courses of treatment may continue study treatment at the discretion of the investigator. Patients discontinuing docetaxel due to toxicity may continue treatment with thalidomide at the discretion of the investigator.

Quality of life is assessed at baseline, before each treatment course, after completion of study treatment, and then every 3 months thereafter.

After completion of study treatment, patients are followed every 3 months for survival.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer, meeting 1 of the following stage criteria:

  * Stage IIIB (with pleural effusion)
  * Stage IIIA or IIIB

    * Previously treated and not eligible for surgery or definitive thoracic radiotherapy
  * Stage IV
* Measurable or evaluable disease
* Documented disease progression during or after standard first-line chemotherapy that may have included taxane
* No untreated brain metastases

  * Patients with previously treated brain metastases are eligible provided they have recovered from prior treatment

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin normal
* SGOT and/or SGPT ≤ 2.5 times upper limit of normal (ULN) AND alkaline phosphatase normal OR
* SGOT and/or SGPT normal AND alkaline phosphatase ≤ 4 times ULN AND no ascites
* Albumin > 3.0 g/dL

Renal

* Creatinine < 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception for 4 weeks before, during, and for ≥ 4 weeks after completion of study treatment
* No HIV positivity
* No peripheral neuropathy > grade 1
* No other malignancy within the past 5 years except inactive nonmelanoma skin cancer or carcinoma in situ of the cervix or breast
* No active infections
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No more than 1 prior systemic chemotherapy regimen for locally advanced or metastatic disease

  * Prior neoadjuvant or adjuvant systemic chemotherapy allowed
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* Recovered from prior radiotherapy

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Complete and partial response rates

SECONDARY OUTCOMES:
Toxicity
Response duration
Survival
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Gillenwater, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States